CLINICAL TRIAL: NCT07193342
Title: Comparison of Computer Controlled Automatic Injection Versus Conventional Injection Regarding Pain ,Anxiety and Child Behavior: "A Randomized Controlled Trial "
Brief Title: Effect of Computer-controlled vs. Conventional Injection on Pain and Anxiety in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Nouran Negm ElDin Mahmoud, Master student, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEDI_INJ_TRIAL2025
Record Dates: First submitted 2025-08-17; First posted 2025-09-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Dental Pain, Dental Anxiety and Child Behavior Are Assess in Response to Dental Injection
Keywords: dental pain; behavior management; local anesthesia in children; pediatric dentistry
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer controlled automatic injection ( Star pen® system) (Experimental): Children will receive local anesthesia using a computer-controlled delivery system (Star Pen® device).
  Interventions: Procedure: computer controlled automatic injection (Star pen® system)
- conventional anesthetic syringe (Active Comparator): Children will receive local anesthesia using a conventional dental syringe.
  Interventions: Procedure: conventional anesthetic syringe

INTERVENTIONS:
Procedure: computer controlled automatic injection (Star pen® system) — local anesthesia will be administered using computer controlled automatic injection(Star pen® system ) to provide slow and consistent anesthetic flow, aiming to reduce pain and anxiety during pediatric dental treatment.
  Arms: computer controlled automatic injection ( Star pen® system)
Procedure: conventional anesthetic syringe — local anesthesia will be administered using a standard manual dental syringe , following conventional injection techniques for pediatric dental patients.
  Arms: conventional anesthetic syringe

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of Computer-Controlled automatic injection device versus conventional injection techniques in pediatric dental patients. The study evaluates differences in pain perception, Anxiety levels ,and behavioral responses during dental procedures among children. by using validated pain and behavior assessment scales, this trial seeks to determine whether the use of automated injection system can improve the overall dental experience for children

DETAILED DESCRIPTION:
This randomized controlled trial aims to compare the effectiveness of Computer-Controlled automatic injection device versus conventional injection techniques in pediatric dental patients. The study focuses on evaluating and analyzing primary outcome ( pain perception) and secondary outcome ( anxiety levels )

Eligible participants will be healthy children who require dental treatment under local anesthesia. Participants will be randomly assigned to one of two Groups :

Groups A: Will receive The Star pen® system , incorporating battery-powered feedback for controlled pressure.

Group B: will receive conventional anesthetic syringe . pain will be assessed both subjectively using age- appropriate pain rating scales (such as Simplified Faces Pain Scale (S-FPS), and objectively using Sound, Eye, Motor scale .

Anxiety will be evaluated by measuring heart rate (objectively ). Child behavior during the procedure will be monitored and rated using venham's behavior scale.

This study aims to determine whether Star pen® system offers a more comfortable and less anxiety - provoking experience for children compared to the conventional method. The result may guide pediatric dentists in selecting the most suitable delivery technique to improve the dental experience and cooperation in pediatric patients.

ELIGIBILITY:
Inclusion criteria:

* Pediatric patients aged 6-9 years.
* Participants are required to undergo dental procedures requiring local infiltration anesthesia.
* Only cooperative patients (scoring 3 or 4 on the Frankl Behavior Scale).
* No prior dental experiences.
* Patients need maxillary infiltration anesthesia.
* No prior symptoms of abscess.
* Only children with ASA I health status (Free from developmental or systemic disorders).
* Parental consent and child assent required for enrollment.

  - Exclusion criteria:
* Medical conditions or systemic illnesses.
* Psychiatric conditions affecting pain or anxiety evaluation.
* Parental refusal or child unwillingness to participate

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Simplified Faces Pain Scale | Immediately after injection procedure
Sound, eye, motor scale | Starting From point entry of anesthesia till end of injection procedure

SECONDARY OUTCOMES:
pulse oximeter | From sitting of patient on dental chair till the end of the injection procedure
Venham Behavior Rating Scale | Starting From point of entry of anesthesia till end of injection procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared